CLINICAL TRIAL: NCT05625074
Title: The Portuguese National Health Service Reality in Varicose Vein Surgery - a Transversal Study on the Early Postoperative of Superficial Venous Surgery.
Brief Title: National Varicose Vein Study - Portugal
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, João Rocha Neves, Principal Investigator, Universidade do Porto
Other Study IDs: UniversidadePorto
Record Dates: First submitted 2022-10-16; First posted 2022-11-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Chronic Venous Insufficiency
Keywords: Venous Insufficiency; Conventional great vein surgery
MeSH Terms: conditions — Venous Insufficiency

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- CHUP Angiology and Vascular Surgery Service: A transversal study, recruiting consecutive patients undergoing great saphenous vein saphenectomy by stripping technique.
  Evaluation and Qol Questionnaires performed at the 30th day of the postoperative period (acceptable scope - 25 to 45 days)
  Interventions: Procedure: Conventional surgery for great saphenous vein insufficiency
- CHUSJ Angiology and Vascular Surgery Service CHUSJ: A transversal study, recruiting consecutive patients undergoing great saphenous vein saphenectomy by stripping technique.
  Evaluation and Qol Questionnaires performed at the 30th day of the postoperative period (acceptable scope - 25 to 45 days)
  Interventions: Procedure: Conventional surgery for great saphenous vein insufficiency
- CHUC Angiology and Vascular Surgery Service CHUSJ: A transversal study, recruiting consecutive patients undergoing great saphenous vein saphenectomy by stripping technique.
  Evaluation and Qol Questionnaires performed at the 30th day of the postoperative period (acceptable scope - 25 to 45 days)
  Interventions: Procedure: Conventional surgery for great saphenous vein insufficiency

INTERVENTIONS:
Procedure: Conventional surgery for great saphenous vein insufficiency — Arch ligation and stripping of great saphenous vein. Prophilatic anticoagulation - Low molecular weight heparin vs DOACs Antibiotics Non-steoridal anti-inflamatory drugs
  Other Names: Arch ligation and stripping of great saphenous vein

SUMMARY:
The National Varicose Vein Study is a cross-sectional, multicenter, observational study. The primary goal is to evaluate the 30 days outcome of the conventional great saphenous vein surgery (stripping) in the treatment of the symptomatic chronic venous insufficiency, comparing the results of difference Portuguese's health centers, comparing the following variables: thrombo-prophylaxis (pharmacology or mechanic; compliance); antimicrobial prophylaxis; quality of life; medication compliance; complications and work incapacity period.

DETAILED DESCRIPTION:
Chronic venous disease is one of the most prevalent pathologies in the world population. It presents a spectrum of variable manifestations, culminating in the most severe form, active venous ulcer. The clinical evaluation, the study of venous anatomy by echo- Doppler and the indications for surgical treatment are standardized in guidelines. The same applies to the techniques for surgical treatment that, in the long term, present equally satisfactory results. Thus, currently, in the Portuguese national health system, the surgical technique most frequently used is conventional surgery. As for postoperative care, namely thromboprophylaxis regimens, analgesia regimens, there is greater variability in its application between clinics and institutions, which may result in significant differences in postoperative recovery. In this way, we intend to develop an observational, cross-sectional and multicenter study, comparing postoperative care protocols and patient compliance and impact on quality of life, as well as absence from work.

The primary goal is to evaluate the 30 days outcome of the conventional great saphenous vein surgery (stripping) in the treatment of the symptomatic chronic venous insufficiency, comparing the results of difference Portuguese's health centers, comparing the following variables: thrombo-prophylaxis (pharmacology or mechanic; compliance); antimicrobial prophylaxis; quality of life; medication compliance; complications and work incapacity period.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated at CHUP, CHUSJ and CHUC
* Male and female;
* Age over 18 years;
* All clinical presentations (C) included in the CEAP classification system;
* Period from November 2022 onwards;
* Conventional surgical treatment of at least one great saphenous vein;
* Patients treated using the following techniques: arch ligation +/- trunk stripping.

Exclusion Criteria:

* Exclusive or concomitant treatment with endovenous surgery (thermal ablation by laser or radiofrequency…);
* Treatment by conservative conventional surgery of the great saphenous vein (CHIVA, ASVAL);
* Varicose surgery not involving the great saphenous vein;
* Age under 18 years;
* Patients treated in hospital units not covered by the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients submitted to surgical treatment of symptomatic insufficiency of the great saphenous vein by conventional surgery (arch ligation +/- trunk stripping), in the postoperative period between 25 and 45 days, in the hospital centers involved in the study starting in November 2022 onwards, until the desired sample volume is reached (50 patients per center).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacological and/or mechanical thromboprophylaxis | In the postoperative period between 25 and 45 days
  Regimen (low molecular weight Heparin vs direct oral anticoagulant; elastic stockings). duration of the thromboprophilaxis regimen
Antibiotic prophylaxis regimens | In the postoperative period between 25 to 45 days
  Duration of the regimen. Beta lactamic vs remaining antibiotics
Impact on quality of Life; | In the postoperative period between 25 to 45 days
  Eq5D5L; 5-level EQ-5D version (EQ-5D-5L)
Impact on quality of Life; | In the postoperative period between 25 to 45 days
  CIVIQ14 - ChronIc Venous Insufficiency QOL Questionnaire (CIVIQ)
Impact on quality of Life; | In the postoperative period between 25 to 45 days
  rVCSS - revised venous clinical seveity score
Compliance with drug therapy; | In the postoperative period between 25 and 45 days
  How many days were recomended to take the drug; How many days the patient took the drug
Complications and extraordinary recourse to health care | In the postoperative period between 25 and 45 days
  Observation in the outpatient clinic and urgency department

SECONDARY OUTCOMES:
Period of work disability | In the postoperative period between 25 and 45 days
  measured in days

CONTACTS AND LOCATIONS:
Locations (1):
- Faculdade de Medicina da Universidade do Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Maeseneer MG, Kakkos SK, Aherne T, Baekgaard N, Black S, Blomgren L, Giannoukas A, Gohel M, de Graaf R, Hamel-Desnos C, Jawien A, Jaworucka-Kaczorowska A, Lattimer CR, Mosti G, Noppeney T, van Rijn MJ, Stansby G, Esvs Guidelines Committee, Kolh P, Bastos Goncalves F, Chakfe N, Coscas R, de Borst GJ, Dias NV, Hinchliffe RJ, Koncar IB, Lindholt JS, Trimarchi S, Tulamo R, Twine CP, Vermassen F, Wanhainen A, Document Reviewers, Bjorck M, Labropoulos N, Lurie F, Mansilha A, Nyamekye IK, Ramirez Ortega M, Ulloa JH, Urbanek T, van Rij AM, Vuylsteke ME. Editor's Choice - European Society for Vascular Surgery (ESVS) 2022 Clinical Practice Guidelines on the Management of Chronic Venous Disease of the Lower Limbs. Eur J Vasc Endovasc Surg. 2022 Feb;63(2):184-267. doi: 10.1016/j.ejvs.2021.12.024. Epub 2022 Jan 11. No abstract available. PMID 35027279
- [Background] O'Donnell TF, Balk EM, Dermody M, Tangney E, Iafrati MD. Recurrence of varicose veins after endovenous ablation of the great saphenous vein in randomized trials. J Vasc Surg Venous Lymphat Disord. 2016 Jan;4(1):97-105. doi: 10.1016/j.jvsv.2014.11.004. Epub 2015 Apr 11. PMID 26946904
- [Background] Brand FN, Dannenberg AL, Abbott RD, Kannel WB. The epidemiology of varicose veins: the Framingham Study. Am J Prev Med. 1988 Mar-Apr;4(2):96-101. PMID 3395496
- [Background] Lurie F, Passman M, Meisner M, Dalsing M, Masuda E, Welch H, Bush RL, Blebea J, Carpentier PH, De Maeseneer M, Gasparis A, Labropoulos N, Marston WA, Rafetto J, Santiago F, Shortell C, Uhl JF, Urbanek T, van Rij A, Eklof B, Gloviczki P, Kistner R, Lawrence P, Moneta G, Padberg F, Perrin M, Wakefield T. The 2020 update of the CEAP classification system and reporting standards. J Vasc Surg Venous Lymphat Disord. 2020 May;8(3):342-352. doi: 10.1016/j.jvsv.2019.12.075. Epub 2020 Feb 27. PMID 32113854